CLINICAL TRIAL: NCT03056469
Title: Patient-Reported Outcomes Integrated in the Follow-up of Patients With Hematological Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REG-72-2016
Record Dates: First submitted 2017-01-25; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Hematological Cancer
Keywords: patient-reported outcomes; supportive care; clinical practice; hematological cancer
MeSH Terms: interventions — prolyl-proline; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: In one randomization arm the participants submit patient-reported outcomes, and the care providers have access to the patient-reported outcomes. In another randomization arm the participants submit patient-reported outcomes, but the care providers do not have access to the patient-reported outcomes. In the last randomization arm the participants are randomized to standard follow-up, do not complete PRO questionnaires and are thus controls.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Care providers do have access to PROs (Active Comparator): Participants complete patient-reported outcome (PRO) questionnaires. Care providers do have access to the PROs and use them in clinical decision making.
  Interventions: Other: Completion of patient-reported outcome (PRO) questionnaires
- Care providers do not have access to PROs (Active Comparator): The participants complete patient-reported outcome (PRO) questionnaires. Care providers do not have access to the PROs.
  Interventions: Other: Completion of patient-reported outcome (PRO) questionnaires
- Control group (No Intervention): Standard follow-up. The participants do not complete PRO questionnaires.

INTERVENTIONS:
Other: Completion of patient-reported outcome (PRO) questionnaires — Patient-reported outcome (PRO) questionnaires are completed at home within one week before a patient-physician consultation at the outpatient clinic. The questionnaires are submitted online or on paper depending on the participants choice.
  Arms: Care providers do have access to PROs; Care providers do not have access to PROs

SUMMARY:
This study investigates if integration of patient-reported outcomes in the follow-up of patients with newly diagnosed, not curable, chronic hematological cancer changes the number and kind of supportive care interventions. Furthermore, this study investigates if the patients feel that they are more involved in a positive way when patient-reported outcomes are integrated in the follow-up of their cancer.

DETAILED DESCRIPTION:
This is a multimethod study. It has a quantitative and a qualitative part. The patient-reported outcome questionnaire European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ C-30) and the patient-reported outcome and patient-reported experience questionnaire The Outcomes and Experiences Questionnaire (OEQ) are completed by the included patients within one week before a patient-physician consultation at the outpatient clinic at one single department of hematology. Baseline is different for different patient groups; 1) for participants receiving a primary treatment baseline is defined as the first patient-physician consultation after the primary treatment ended, 2) for patients continuously receiving medical treatment baseline is defined as the first patient-physician consultation after starting medical treatment, and 3) for patients followed using a watch and wait strategy baseline is defined as the first patient-physician consultation after deciding the watch and wait strategy. Each patient completes the questionnaires for 2 years. The questionnaires can be completed online or on paper depending on the patients choice. Answers from both questionnaires are eligible to all health care professionals in the outpatient clinic in an internet-based tool. A summary of scores from the EORTC QLQ C-30, and the answers and the score from the OEQ, are written in the medical record.

This study investigates, if use of the patient-reported outcome (PRO) questionnaires are useful in the assessment of the patients needs and health care providers decision making regarding supportive care interventions. It investigates, if completion of PRO questionnaires changes the number and kind of supportive care interventions.

Observations of patient-physician consultations and individual interviews with patients are used to capture the impact of the questionnaires on the consultations and patients evaluation of the use of the questionnaires.

This study also investigates, if patients completion of PRO questionnaires and health care professionals use of the questionnaires in clinical decision making changes the number of contacts between patients and a department of hematology and the number of paraclinical interventions.

ELIGIBILITY:
Inclusion Criteria:

* patients newly diagnosed with not curable, chronic hematological cancer
* ≥18 years old
* oral and written informed consent

Exclusion Criteria:

* participation in another intervention study
* psychological or physiological conditions that may prevent compliance/adherence to the study
* patients do not wish to be included in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-03 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Supportive care interventions | Three and a half year
  Number and kind of supportive care interventions are registered. Supportive care actions are defined as: a) a plan for rehabilitation, b) an intervention by a physiotherapist, occupational therapist, dietician, or social worker, c) consultation with a psychologist or talk with a priest, d) an intervention done by a general practitioner because of the hematological cancer after contact between the hematological department and the general practitioner, e) use of offers like group talks etc offered by the Danish Cancer Society, or f) other supportive care interventions

SECONDARY OUTCOMES:
Patients satisfaction with the interventions done by a department of hematology | Three and a half year
  Patients satisfaction with the interventions done by a department of hematology are measured using a patient-reported experience questionnaire
Impact of the use of PRO questionnaires on the consultation and patient satisfaction with and evaluation of the use of patient-reported outcomes in the outpatient clinic | Three and a half year
  The impact of the use of PRO questionnaires on the consultation and patients satisfaction with and evaluation of the use of patient-reported outcomes in the outpatient clinic are investigated by observation of conversations between doctors and patients in the outpatient clinic, and furthermore investigated by individual interviews
Contacts to the outpatient clinic at department of hematology | Three and a half year
  All contacts between the patients and the department of hematology are registered. Are there more/less/equal number and kind of contacts to the outpatient clinic at department of hematology when using patient-reported outcomes compared to when not using patient-reported outcomes?
Paraclinical interventions | Three and a half year
  All paraclinical actions ordered by the department of hematology are registered. Are more/less/equal number and kind of paraclinical interventions done when using patient-reported outcomes compared to when not using patient-reported outcomes?

CONTACTS AND LOCATIONS:
Overall Officials: Hans Hasselbalch, professor, Study Chair — Department of Hematology, Zealand University Hospital, Vestermarksvej 9, 4000 Roskilde, Denmark
Locations (1):
- Department of Hematology, Zealand University Hospital, Roskilde, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thestrup Hansen S, Kjerholt M, Friis Christensen S, Brodersen J, Holge-Hazelton B. Nurses' Experiences When Introducing Patient-Reported Outcome Measures in an Outpatient Clinic: An Interpretive Description Study. Cancer Nurs. 2021 Mar-Apr 01;44(2):E108-E120. doi: 10.1097/NCC.0000000000000808. PMID 32217877